CLINICAL TRIAL: NCT01069198
Title: A Randomized, Double Blind, Community Trial to Assess the Efficacy of a Combination of Anti-helminth, and Vitamin A, Zinc and Iron Supplementation in Preventing Visceral Leishmaniasis (VL) Disease Among Asymptomatic Individuals With VL
Brief Title: A Community Trial for Visceral Leishmaniasis (VL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Access to Advanced Health Institute (AAHI) (Other); Nagasaki University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-09018
Record Dates: First submitted 2010-02-14; First posted 2010-02-17 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2010-01

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; Kala-azar; Bangladesh; Malnutrition; Asymptomatic; Albendazole; Iron; Zinc; Vitamin A
MeSH Terms: conditions — Leishmaniasis, Visceral; Malnutrition | interventions — Albendazole; Iron; Zinc; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: Albendazole, Iron, Zinc and Vitamin A
- Non-intervention group (Placebo Comparator): Non-intervention group will receive placebo following the same schedule as intervention group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Albendazole, Iron, Zinc and Vitamin A — single oral dose of 200,000 IU Vitamin A at baseline and after six months, 35 mg and 65 oral elemental iron for subject aged <5 and >=5 years respectively everyday for two months starting from enrollment; 10 mg oral zinc for 10 consecutive days each month for 6 months; and a single 400 mg oral dose of albendazole at 3-months' intervals.
  Arms: Intervention group
Other: Placebo — Placebo
  Arms: Non-intervention group

SUMMARY:
Visceral leishmaniasis (VL) / Kala-azar (KA) is a public health problem in the many countries in the world including Bangladesh. Where more than 90,000 VL cases have been reported since 1994. The disease is fatal if not treated. Even with treatment the mortality rate is high (10%). VL is a vector-borne disease, caused by the parasite Leishmania donovani (LD) and is transmitted by female sandfly sp. Phlebotomus argentipes. Not all people exposed to the LD parasite develop disease. According to our observation only about 30% of the infected with LD parasite develop disease within one year of diagnosis. Malnutrition and intestinal helminth infection have been found to be associated with the risk of active VL. Down regulation of Th1 cellular immune response confers susceptibility to active VL. Both malnutrition and intestinal helminth infection down regulate the Th1 cellular immune response. Till now there is no established prophylaxis against active VL among the people exposed to the LD infection. Many studies including ours have been shown that periodic regular deworming reduced malnutrition significantly. Micronutrient such as zinc and iron as well vitamin A supplementation also improve malnutrition and may enhance Th1 cellular immune response. Thus we hypothesize that periodic deworming and. micronutrient and vitamin A supplementation together may reduce the risk of active VL among the people exposed to the LD infection.

The study will be carried out in the Harirampur union, Trishal, Mymensingh. This area is highly endemic for VL. Two hundred asymptomatic VL patients aged 2-60 will be enrolled to the study. Children aged less than 2 years, pregnant women, active VL case, person with chronic disease, disable individuals and those who will refuse written consent will not be enrolled to the study. After enrollment subjects will be divided into two groups through randomization. One group will receive deworming and nutritional supplement (intervention group) and other group will receive placebo (placebo group). Two groups will be followed for 12 months through active surveillance for developing of active VL. In addition morbidity data, monthly stool sampling, monthly anthropometry, urine and blood sampling at baseline, before and after treatment of active VL will be carried out Successful completion of the study and derived results from it will provide useful information that whether periodic deworming with micronutrient and vitamin A supplementation can reduce the risk of active VL among the people exposed to the LD infection.

ELIGIBILITY:
Inclusion Criteria:

* An individual with positive rK39 strip test, without past history of VL and/or symptom and sign of chronic illness.

Exclusion Criteria:

* Children aged < 2 years,
* Adults aged > 60 years,
* Patients of active VL,
* Pregnant women,
* People with chronic or debilitating conditions.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of deworming and supplementation with iron, zinc and vitamin A on incidence of active VL among the individuals with asymptomatic VL. | 12 months

SECONDARY OUTCOMES:
To investigate the prevalence of asymptomatic and symptomatic VL among the households with a past case of VL. To measure the parasite load in the blood by Real Time PCR and to study the association of blood parasite load with active VL. | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - International Centre For Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh
  - International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka